CLINICAL TRIAL: NCT05610644
Title: Impact of Time Restricted Feeding on Daily Protein Requirements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 275081
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Nutrition Disorders in Old Age

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TRF of RDA (Active Comparator): A time-restricted model of consumption of the RDA of protein/day.
  Interventions: Other: isocaloric, isonitrogenous meals
- TRAD of RDA (Active Comparator): A typical American dietary ingestion pattern of the RDA of protein/day.
  Interventions: Other: isocaloric, isonitrogenous meals
- TRF of 2RDA (Experimental): A time-restricted model of consumption of twice the RDA of protein/day.
  Interventions: Other: isocaloric, isonitrogenous meals
- TRAD of 2RDA (Experimental): A typical American dietary ingestion pattern of twice the RDA of protein/day.
  Interventions: Other: isocaloric, isonitrogenous meals

INTERVENTIONS:
Other: isocaloric, isonitrogenous meals — Participants will eat prepared study meals for 3 days that have either the RDA of protein per day or twice the RDA of protein per day.

SUMMARY:
The investigators aim to assess 24-hour protein kinetics at two different levels of protein intake: 0.8 (RDA) and 1.6g/kg/day (2RDA) during a normal dietary (TRAD) and a time restricted feeding (TRF) pattern in older adults.

DETAILED DESCRIPTION:
The investigators aim to assess 24-hour protein kinetics at two different levels of protein intake: 0.8 (RDA) and 1.6g/kg/day (2RDA) during a normal dietary (TRAD) and a time restricted feeding (TRF) pattern in older adults. Individuals in the TRF pattern will only consume food during a 6-hour eating period and fast for the remaining 18 hours. Individuals in the TRAD pattern will consume isocaloric and isonitrogenous (RDA or 2RDA) diet but consume an all-beef-breakfast. Participants will consume oral stable isotopes to measure muscle protein synthesis (MPS), whole-body muscle protein breakdown (MPB), and whole-body protein balance (WBPB). Appropriate muscle, blood samples, and urine will be collected throughout a 24-hour metabolic trial following a 2-day controlled diet.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 50-75 years.
2. BMI 20-30 kg/m2 inclusive.
3. Capable of providing informed consent.
4. COVID-19 negative and/or asymptomatic

Exclusion Criteria:

1. Subject who does not/will not eat animal protein sources.
2. Body mass index <20 or >30.
3. Hemoglobin <10g/dL at screening.
4. Platelets <150,000/uL at screening.
5. History of diabetes.
6. History of chemotherapy or radiation therapy for cancer in the 6 months prior to enrollment.
7. History of gastrointestinal bypass/reduction surgery.
8. History of a chronic inflammatory disease (e.g. what?)
9. Currently receiving androgen (e.g., testosterone) or anabolic (e.g., GH, IGF-I) therapy.
10. Currently using prescription blood thinning medications.
11. Currently using corticosteroid medications.
12. Unable or unwilling to suspend aspirin use for 7 days prior to Visit 3.
13. Unwilling to avoid using protein or amino-acid supplements during participation.
14. Subjects who are unwilling to fast overnight.
15. Participating in >200 minutes/week of vigorous exercise and/or >4 days/week of resistance training.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Whole-body protein balance | 24 hours
  Volume of net protein produced per unit of time

CONTACTS AND LOCATIONS:
Overall Officials: David Church, Principal Investigator — UAMS (University of Arkansas for Medical Sciences)
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No